CLINICAL TRIAL: NCT01811342
Title: Evaluation of the Masimo Continuous Hemoglobin Monitor With Polar Plot Methodology
Brief Title: Continuous Hemoglobin Evaluation
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 348788
Record Dates: First submitted 2013-03-07; First posted 2013-03-14 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Anemia
Keywords: Hemoglobin; Patient Monitoring
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemoglobin Measurement: Patients requiring intra-operative hemoglobin measurement.

SUMMARY:
Evaluate potential sources of error that affect the accuracy of continuous hemoglobin monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgery.

Exclusion Criteria:

* 0

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Masimo Continuous Hemoglobin Monitor with Polar Plot Methodology | One year
  Determine the influence of initial calibration and intraoperative oxygenation variables on the correlation between SpHgb and clinical values

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States